CLINICAL TRIAL: NCT02586649
Title: A Randomized, Double-blind, Placebo-controlled Trial to Determine the Effects and Duration of Action of Tiotropium Bromide on Pulmonary Function in Persons With SCI
Brief Title: 24hr Effects of Tiotropium Bromide in Tetraplegia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Gregory Schilero, Director of Sleep Lab/ICU, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SCH-14-019
Record Dates: First submitted 2015-10-13; First posted 2015-10-26 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury
Keywords: tiotropium bromide
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Tiotropium Bromide; Cholinergic Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tiotropium Bromide group (Experimental): The study participants will be randomly assigned to receive Tiotropium bromide,single dose (inhalation capsule - 18 mcg) over the course of 24 hours on day one of visit 1 or during visit 3.On the day of the first scheduled visit ( visit 1 ),study participants will be asked to arrive between 12-1 pm at the pulmonary laboratory at the JJPVAMC (7A-13). Baseline blood pressure (BP) and heart rate (HR) measurements will be obtained prior to drug administration. Tiotropium bromide capsule containing active ingredients will be orally inhaled through a SPIRIVA HandiHaler. Measurements of exhaled nitric oxide, pulmonary function ( spirometry , static lung volumes and specific airway conductance) will be performed at 20 and 24 hours. The same schedule will be followed for visits 3 and 4;vists 3 and 4 will be scheduled between 14 and 21 days after visit 2.
  Interventions: Drug: Tiotropium Bromide; Drug: Placebo
- Placebo (Placebo Comparator): The study participants will be randomly assigned to receive placebo , single dose (inhalation capsule - 18 mcg) over the course of 24 hours on day one of visit 1 or during visit 3.On the day of the first scheduled visit ( visit 1 ),study participants will be asked to arrive between 12-1 pm at the pulmonary laboratory at the JJPVAMC (7A-13). Baseline blood pressure (BP) and heart rate (HR) measurements will be obtained prior to drug administration. Placebo capsule containing active ingredients will be orally inhaled through a SPIRIVA HandiHaler. Measurements of exhaled nitric oxide, pulmonary function ( spirometry , static lung volumes and specific airway conductance) will be performed at 20 and 24 hours. The same schedule will be followed for visits 3 and 4;vists 3 and 4 will be scheduled between 14 and 21 days after visit 2.
  Interventions: Drug: Tiotropium Bromide; Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium Bromide — Tiotropium bromide is an anticholinergic used to study bronchodilatation and improvement of pulmonary function in tetraplegic patients
  Other Names: Anticholinergic
Drug: Placebo — Placebo is a non-active inhalation capsule .

SUMMARY:
Respiratory complications are the leading cause of death during the initial year after acute SCI, and the third leading cause of death thereafter. Complete or partial loss of respiratory muscle innervations in individuals with cervical and high thoracic injuries leads to inadequate ventilation and inability to effectively clear secretions, often prompting supportive ventilation following initial injury. Development of atelactasis, pneumonias and respiratory failure are the most common respiratory complications observed during the acute phase of injury. It is well known that a restrictive ventilatory defect, dependent upon the level and completeness of injury, is apparent in individuals with chronic cervical SCI. Respiratory functional impairment might be further compromised in these individuals, the majority of whom share many aspects of obstructive airway physiology commonly associated with asthma. The asthma-like features that individuals with chronic cervical SCI demonstrate have been hypothesized to be due to overriding cholinergic airway tone carried by intact vagal (parasympathetic) nerve fibers arising from the brainstem, whereas sympathetic innervations is interrupted at the level of the upper thoracic spinal cord. Whether airway narrowing and AHR in chronic cervical SCI is also related to chronic airway inflammation is unknown, although it is conceivable that repeated respiratory infections or, possibly, a neurogenic component, could contribute to chronic airway inflammation.

Therefore, the investigators aim to assess how long-acting bronchodilator (tiotropium bromide) affects various indices of lung function, including: pulmonary function tests, levels of inflammation and cough strength across 24 hours after receiving study drug. Results will be analyzed for baseline, 1 hour, 3 hours, 20 hours and 24 hours post drug inhalation for both active medication and non-active placebo.

DETAILED DESCRIPTION:
In addition to a restrictive ventilatory defect stemming for respiratory muscle paralysis, cervical SCI (tetraplegia) is associated with obstructive airway physiology similar to that associated with asthma. The investigators hypothesize that these aspects of obstructive physiology stem from unopposed increases in cholinergic airway tone as a result of autonomic imbalance; where vagal innervation (cholinergic neurotransmission) to the lungs is intact, and the bronchodilating adrenergic influences of sympathetic pathways are interrupted. The investigators demonstrated using spirometric criteria, significant bronchodilator responses in approximately 50% of subjects with tetraplegia following inhalation of short acting beta-2 agonists (albuterol sulfate) and anticholinergic agents (ipratropium bromide). When specific airway conductance (sGaw), a more sensitive indicator of bronchodilation, was assessed via whole body plethysmography, significant bronchodilation and restoration of normal airway caliber was noted in all subjects.

Intuitively, one might expect that through bronchodilation susceptible individuals with tetraplegia who already have compromised respiratory muscle strength and weakened cough might benefit from better airway clearance, and via increases in lung volumes improve the length-tension relationship of residual expiratory muscles for initiation of more forceful coughs. Based upon a comparative study of the bronchodilator effects of ipratropium bromide versus albuterol in persons with tetraplegia (in publication), it appears that ipratropium bromide elicited greater bronchodilation, perhaps because of the specificity of action in blocking acetylcholine binding to the muscarinic-3 (M3) airway smooth muscle receptor. The investigators purpose in this preliminary study is to assess whether salutary effects upon pulmonary function, cough strength, and airway inflammation are observed across a twenty-four hour period following inhalation of a single dose of tiotropium bromide 18 mcg inhalational capsule versus placebo utilizing a double-blind crossover design in persons with chronic stable tetraplegia.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Spinal Cord Injury (>1 year post-injury)
2. Stable tetraplegia (level of injury C3-C8, non-ventilator dependent)
3. Male or female between the ages 18-65

Exclusion Criteria:

1. Smoking, active or history of smoking during last 6 months;
2. Ventilator dependent;
3. Known history of asthma, COPD or inflammatory disease during lifetime;
4. Active or recent (within 3 months) respiratory infection;
5. Use of medications known to affect the respiratory system;
6. Use of medications known to alter airway caliber
7. Uncontrolled hypertension;
8. Glaucoma or cataracts;
9. History of milk protein allergy
10. Pregnant or trying to become pregnant
11. Lack of mental capacity to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Spirometry values from baseline | Baseline,one hours post,three hours post,twenty hours post,twenty four hours post
  During Visit 1 (0,1 and 3 hours post-drug); Visit 2 (20 and 24 hours post-drug); Visit 3( between 14 and 21 days after visit 2- 0,1 and 3 hours post-drug); Visit 4 (following visit 3)
Change in Exhaled Nitric Oxide ( FeNO ) | Baseline,one hours post,three hours post,twenty hours post,twenty four hours post
  During Visit 1 (0,1 and 3 hours post-drug); Visit 2 (20 and 24 hours post-drug); Visit 3( between 14 and 21 days after visit 2- 0,1 and 3 hours post-drug); Visit 4 (following visit 3)

SECONDARY OUTCOMES:
Change in Lung volumes ( Plethysmography ) | Baseline,one hours post,three hours post,twenty hours post,twenty four hours post
  During Visit 1 (0,1 and 3 hours post-drug); Visit 2 (20 and 24 hours post-drug); Visit 3( between 14 and 21 days after visit 2- 0,1 and 3 hours post-drug); Visit 4 (following visit 3)
Change in Airway Resistance by Impulse Oscillometry System (IOS) | Baseline,one hours post,three hours post,twenty hours post,twenty four hours post
  During Visit 1 (0,1 and 3 hours post-drug); Visit 2 (20 and 24 hours post-drug); Visit 3( between 14 and 21 days after visit 2- 0,1 and 3 hours post-drug); Visit 4 (following visit 3)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Schilero, MD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J Peters VA Medical Center, New York, New York, United States

REFERENCES:
- [Background] Radulovic M, Schilero GJ, Wecht JM, La Fountaine M, Rosado-Rivera D, Bauman WA. Exhaled nitric oxide levels are elevated in persons with tetraplegia and comparable to that in mild asthmatics. Lung. 2010 Jun;188(3):259-62. doi: 10.1007/s00408-009-9207-x. Epub 2009 Dec 15. PMID 20012982
- [Result] DeVivo MJ, Krause JS, Lammertse DP. Recent trends in mortality and causes of death among persons with spinal cord injury. Arch Phys Med Rehabil. 1999 Nov;80(11):1411-9. doi: 10.1016/s0003-9993(99)90252-6. PMID 10569435
- [Result] Spungen AM, Dicpinigaitis PV, Almenoff PL, Bauman WA. Pulmonary obstruction in individuals with cervical spinal cord lesions unmasked by bronchodilator administration. Paraplegia. 1993 Jun;31(6):404-7. doi: 10.1038/sc.1993.67. PMID 8337005
- [Result] Almenoff PL, Alexander LR, Spungen AM, Lesser MD, Bauman WA. Bronchodilatory effects of ipratropium bromide in patients with tetraplegia. Paraplegia. 1995 May;33(5):274-7. doi: 10.1038/sc.1995.62. PMID 7630654
- [Result] Sikka N, Margolis G. Understanding diversity among prehospital care delivery systems around the world. Emerg Med Clin North Am. 2005 Feb;23(1):99-114. doi: 10.1016/j.emc.2004.09.007. PMID 15663976